CLINICAL TRIAL: NCT05413109
Title: COMPression of Left Main coRonary artEry in patientS With Pulmonary Arterial Hypertension aSymptomatIc fOr aNgina
Acronym: COMPRESSION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COMPRESSION
Record Dates: First submitted 2022-06-07; First posted 2022-06-09 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coronary-CT (Experimental): Patients with PAH, asymptomatic for angina, with a PA trunk diameter ≥ 4 cm that undergo a coronary-CT scan examination
  Interventions: Radiation: Coronary CT angiography

INTERVENTIONS:
Radiation: Coronary CT angiography — A coronary CT angiography will be used to study the relationship between the PA and the LMCA and 4 radiological patterns will be considered:
  1. "Normal": minimum distance between the two vessels> 1 mm;
  2. "Proximity": distance between the two vessels ≤1 mm without displacement or stenosis of the LMCA;
  3. "Dislocation": dislocation of the LMCA by the main branch of the PA with a take-off angle <60 ° (the take-off angle is defined by the angle formed by the perpendicular to the aortic valve ring and the longitudinal axis of the LMCA);
  4. "Compression": stenosis of the LMCA ≥50% due to extrinsic compression by the PA.

SUMMARY:
The prevalence of critical ab extrinsic compression of left main coronary artery (LMCA) is very high in patients with pulmonary arterial hypertension (PAH) symptomatic for angina (up to 40% according to a recent study of 121 patients with PAH). The element that most of all correlates with the degree of coronary stenosis is the diameter of the pulmonary artery (PA). In particular, a diameter ≥ 40 mm has a sensitivity of 83% and a specificity of 70% in patients with angina. Critical stenosis of LMCA is a risk factor for sudden death and in these condition percutaneous coronary angioplasty with stent implantation has proven to be a safe and effective long-term procedure. Preliminary data from a retrospective analysis of the registry of patients with PAH in Bologna (ARCA registry, 109/2016/U/Oss) highlights that even in PAH patients asymptomatic for angina, compression of LMCA can occur in up to 13% of patients and the main predictive parameter of compression was found to be a diameter ≥ 42 mm (with a sensitivity of 87% and a specificity of 77%). Performing a screening test by coronary-CT scan in all subjects suffering of PAH with a PA diameter ≥ 40 mm even if asymptomatic for angina could therefore help to identify patients with PAH at increased risk for sudden death at an early stage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PAH (group 1 of World Health Organization pulmonary hypertension classification) who have undergone at least one pulmonary CT angiography with a PA trunk diameter ≥ 4 cm
* Age ≥18 years
* Asymptomaticity for angina pectoris or anginal equivalent

Exclusion Criteria:

* Severe chronic kidney disease [Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) estimated glomerular filtration rate <30 ml/min) or need for dialysis
* Major allergy to iodinated contrast agent
* Intolerance or allergy to acetylsalicylic acid or clopidogrel
* History of stroke or transient ischemic attack in the last 6 months or a history of intracranial haemorrhage
* Known cerebral arteriovenous malformation or aneurysm
* Known moderate or severe hepatic insufficiency (Child Pugh B or C)
* Thrombocytopenia (<100.000/μL) or anemia (hemoglobin <10 g/dL)
* Active bleeding or factors which, in the investigator's judgment, significantly increase the risk of bleeding
* Major surgery in the past 30 days
* Cancer in the active phase
* Pregnancy or breastfeeding
* Patient prognosis <1 year in the opinion of the investigator
* Any condition that increases the risk of non-compliance or of being lost to follow-up
* Patients who have already undergone a LMCA angioplasty
* Failure to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of extrinsic compression of the LMCA | Baseline
  To evaluate the incidence of extrinsic compression of the LMCA in patients with PAH and a PA diameter of at least 4 cm, asymptomatic for angina pectoris, subjected to a screening test by coronary CT angiography

SECONDARY OUTCOMES:
Incidence of extrinsic compression of the LMCA by radiological pattern | Baseline
  To evaluate the incidence of extrinsic compression of LMCA in the different possible radiological patterns described by coronary CT angiography (compression, dislocation, contiguity)
Number of participants undergoing LMCA angioplasty with in-hospital complications | Baseline, 1 year
  To evaluate the safety of the LMCA angioplasty in patients with LMCA critical ab extrinsic compression by evaluating the incidence of in-hospital complications [death, myocardial infarction, transient ischemic attack (TIA) or stroke, re-angioplasty, or acute stent thrombosis, vascular complications, acute kidney injury] and at 1 year [death, myocardial infarction, TIA or stroke, restenosis, stent thrombosis and bleeding whose severity will be assessed according to the Bleeding Academic Research Consortium (BARC) classification]
Six minute walking test (6MWT) | Baseline, 6 months
  In patients who will undergo LMCA angioplasty for LMCA critical ab extrinsic compression the change from baseline in the six-minute walk test (6MWT) after the procedure will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Dardi, PhD, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna (Italy)
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galie N, Saia F, Palazzini M, Manes A, Russo V, Bacchi Reggiani ML, Dall'Ara G, Monti E, Dardi F, Albini A, Rinaldi A, Gotti E, Taglieri N, Marrozzini C, Lovato L, Zompatori M, Marzocchi A. Left Main Coronary Artery Compression in Patients With Pulmonary Arterial Hypertension and Angina. J Am Coll Cardiol. 2017 Jun 13;69(23):2808-2817. doi: 10.1016/j.jacc.2017.03.597. PMID 28595696
- [Background] Saia F, Palazzini M, Taglieri N, Manes A, Dardi F, Rinaldi A, Gotti E, Galie N. Reply: Left Main Extrinsic Compression in Pulmonary Arterial Hypertension: From Identification to Percutaneous Coronary Intervention Optimization. J Am Coll Cardiol. 2017 Nov 7;70(19):2460-2461. doi: 10.1016/j.jacc.2017.08.067. No abstract available. PMID 29096819
- [Background] Saia F, Dall'Ara G, Marzocchi A, Dardi F, Palazzini M, Manes A, Taglieri N, Marrozzini C, Rinaldi A, Galie N. Left Main Coronary Artery Extrinsic Compression in Patients With Pulmonary Arterial Hypertension: Technical Insights and Long-Term Clinical Outcomes After Stenting. JACC Cardiovasc Interv. 2019 Feb 11;12(3):319-321. doi: 10.1016/j.jcin.2018.08.002. No abstract available. PMID 30732740